CLINICAL TRIAL: NCT06171750
Title: A Phase I Open-Label, Dose Escalation Study of the Safety and Tolerability of Tolododekin Alfa (ANK-101) in Advanced Solid Tumors
Brief Title: Phase I Study of Tolododekin Alfa (ANK-101) in Advanced Solid Tumors
Acronym: ANCHOR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ankyra Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANK-101-001
Record Dates: First submitted 2023-11-29; First posted 2023-12-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumor; Cutaneous Tumor; Subcutaneous Tumor; Malignant Solid Tumor; Solid Tumor; Metastatic Solid Tumor; Metastasis to Soft Tissue; Non Small Cell Lung Cancer; Cutaneous Squamous Cell Carcinoma
Keywords: intratumoral; intratumoral injection; solid tumors; superficial tumors; nodal tumors; subcutaneous tumors; visceral tumors
MeSH Terms: conditions — Skin Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- tolododekin alfa (ANK-101) IT Injection in Superficial Lesions (Experimental): IT injections of ANK-101 once every 3 weeks into superficial lesions
  Interventions: Drug: tolododekin alfa
- tolododekin alfa (ANK-101) IT Injection in Visceral Lesions (Experimental): IT injections of ANK-101 once every 3 weeks into visceral lesions and every 6 weeks in the expansion
  Interventions: Drug: tolododekin alfa
- tolododekin alfa (ANK-101) IT Injection in Combination with Cemiplimab (Experimental): IT injections of ANK-101 once every 3 weeks in combination with Cemiplimab into patients with high-risk locally advanced or metastatic CSCC that have superficial lesions
  Interventions: Drug: tolododekin alfa; Drug: Cemiplimab

INTERVENTIONS:
Drug: tolododekin alfa — IT administration of ANK-101 once every 3 weeks for up to 12 weeks (4 doses); if there is no disease progression, decrease in clinical performance status or unacceptable toxicity, participants may receive 4 additional doses of ANK-101.
  Other Names: ANK-101
Drug: Cemiplimab — Participants will receive four cycles of ANK-101 in combination with Cemiplimab. If there is no significant clinical deterioration as determined by the Investigator or unacceptable toxicity at Week 12, participants may receive an additional four cycles of the combination treatment. After stopping ANK-101 treatment, participants may stay on Cemiplimab monotherapy for an additional 24 weeks.
  Other Names: Libtayo
  Arms: tolododekin alfa (ANK-101) IT Injection in Combination with Cemiplimab

SUMMARY:
This is a Phase 1, multicenter, open-label dose escalation study to determine the safety and tolerability of intratumoral (IT) injection of tolododekin alfa (ANK-101) in participants with advanced solid tumors who have progressed during or after receiving standard of care (SOC) therapy or who will not benefit from such therapy. The study will be conducted in three parts; in Part 1, participants with superficial lesions will receive ANK-101 as a single agent; in Part 2, participants with visceral lesions will receive ANK-101 as a single agent; and in Part 3, participants with cutaneous squamous cell carcinoma (CSCC) will receive ANK-101 in combination with cemiplimab.

DETAILED DESCRIPTION:
This Phase 1 first-in-human (FIH) study will: 1) evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic effects and preliminary clinical activity of tolododekin alfa (ANK-101) administered as an intratumoral (IT) injection in participants with superficial or visceral lesions; 2) determine the recommended dose for expansion (RDE) of ANK-101; and 3) to determine the safety and tolerability of ANK-101 in combination with cemiplimab.

For parts 1 and 2, the study design consists of six sequential dose-escalation cohorts. Part 1 will enroll participants with advanced solid tumors, with cutaneous, subcutaneous or nodal disease (accessible by clinical palpation or ultrasound guidance). Part 2 will start once the DLT period of dose level 1 in Part 1 is completed and dose level 2 is opened. Part 2 will enroll participants with visceral disease (accessible by interventional radiology or endoscopic techniques). Participants in Part 2 may also have superficial lesions that can be injected if in the Investigator's opinion this is clinically indicated.

Ten participants with non-small cell lung cancer (NSCLC) will be dosed in a Part 2 dose expansion cohort at the RDE.

Part 3 will start once dose escalation for Part 1 is complete and the RDE is identified. Part 3 will consist of ANK-101 in combination with cemiplimab in 15 participants with high-risk locally advanced or metastatic CSCC that have superficial lesions for injection. Participants will be treated with ANK-101 given as IT injections once every three weeks at the RDE in combination with cemiplimab.

Enrollment in Part 3 will include a safety run-in of 5 participants. Following the first dose of the 5th participant, enrollment will pause for 21 days before opening enrollment to the remaining 10 participants or stopping further enrollment.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age on day of signing informed consent
* histologically or cytologically confirmed diagnosis of cutaneous, subcutaneous, soft tissue, or nodal advanced solid tumor malignancy; metastatic disease eligible
* measurable disease per RECIST v1.1 - Note: Must have at least 1 tumor lesion with longest dimension of ≥ 10 mm (≥ 15 mm for the short axis for malignant lymph node lesions) that - For Part 1 only: can be easily palpated or detected by ultrasound to facilitate IT injection of ANK-101 (i.e., tumor in skin, muscle, subcutaneous tissue, or accessible lymph node) or; - For Part 2 only: can be accessed by interventional radiologic or endoscopic procedures for injection (e.g., ultrasound or computed tomography [CT] guided). - For Part 2 Dose Expansion Cohort only: Histologically confirmed Stage III or Stage IV NSCLC
* Part 3 CSCC Combination Cohort: Histologically confirmed high-risk locally advanced or metastatic CSCC not amenable to surgical management as determined by a multidisciplinary tumor board.
* documented disease progression, be refractory to, or intolerant of existing SOC therapy(ies) known to provide clinical benefit (including surgical cure) or not be eligible for SOC therapy(ies)
* ECOG performance status 0-1
* life expectancy > 12 weeks
* adequate bone marrow, hepatic and renal function
* baseline electrocardiogram (EKG) without evidence of acute ischemia or prolonged QTc interval > 460 msec
* Human immunodeficiency virus (HIV) infected participants must be on anti-retroviral therapy (ART) and have well-controlled HIV infection/disease
* last dose of previous anticancer therapy (including investigational agents) ≥ 28 days, radiotherapy ≥ 14 days (targeted palliative radiotherapy is allowed for lesions not planned for injections), or surgical intervention ≥ 21 days prior to the start of treatment
* resolution of all prior anticancer therapy toxicities (except for alopecia or vitiligo) to ≤ Grade 1 (as per NCI CTCAE Version 5.0)
* willing to provide pre- and post-treatment tumor biopsy samples if medically feasible
* participant is capable of understanding and complying with protocol requirements

Exclusion Criteria:

* injectable tumors impinging upon major airways or blood vessels
* prior treatment with recombinant interleukin-12 (IL-12)
* have received systemic therapy with immunosuppressive agents ≤ 28 days before the start of treatment
* have received live vaccines within 28 days prior to the start of ANK-101 treatment
* have primary or acquired immunodeficient states (e.g., leukemia, lymphoma)
* a woman of childbearing potential (WOCBP) who has a positive serum pregnancy test (within 72 hours) prior to the start of treatment or female participant who is breastfeeding
* prior organ transplantation
* known history of hepatitis B virus, known active hepatitis C virus, or a positive serological test at screening within 28 days prior to the start of treatment
* HIV-infected participants with a history of Kaposi sarcoma and/or Multicentric Castleman Disease
* active autoimmune disease or medical conditions requiring chronic steroid (i.e., ≥ 20 mg/day prednisone or equivalent) or other immunosuppressive therapy within 28 days prior to the start of treatment
* known active central nervous system (CNS) metastases
* congestive heart failure (> New York Heart Association Class II), active coronary artery disease, unevaluated new onset angina within 3 months or unstable angina (angina symptoms at rest), or clinically significant cardiac arrhythmias
* uncontrolled bleeding disorders within 4 weeks prior to the start of treatment or known bleeding diathesis - Note: Part 2 only: Participants with active bleeding diathesis or requirement for therapeutic anticoagulation that cannot be interrupted or altered for procedures
* history of hypersensitivity to compounds of similar biological composition to IL-12, aluminum hydroxide, or drugs formulated with polysorbate-20
* other systemic conditions or organ abnormalities that, in the opinion of the Investigator, may interfere with the conduct and/or interpretation of the current study
* any acute or chronic psychiatric problems or substance abuse disorder that, in the opinion of the Investigator, make the participant unsuitable for participation
* Part 3 only: prior Grade 3 or greater immune-mediated adverse events (imAEs) following treatment with an agent that blocks the programmed cell death protein 1 (PD-1)/programmed cell death ligand 1 (PD-L1) pathway.
* Part 3 only: hypersensitivity to cemiplimab or any of its excipients or contraindications to cemiplimab per approved local labeling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and characteristics of DLTs (Parts 1 and 2 only) and TEAEs | From Day 1 to 90 days after last injection of ANK-101
  Number and percentage of participants reporting each DLT or TEAE.
RDE of ANK-101 | Approximately 12 months
  Defined based on the rate of DLTs and TEAEs
Incidence and characteristics of TEAEs of ANK-101 in combination with Cemiplimab according to NCI CTCAE v5.0 (Part 3 only) | From Day 1 to 90 days after last injection of ANK-101 in combination with Cemiplimab.
  Number and percentage of participants reporting each TEAE.

SECONDARY OUTCOMES:
PK: Cmax of IL-12-ABP | Up to 2 years
  PK of IL-12-ABP as assessed by maximum plasma concentration (Cmax)
PK: AUC of IL-12-ABP | Up to 2 years
  PK of IL-12-ABP as assessed by area under the time-concentration curve (AUC)
PK: t ½ of IL-12-ABP | Up to 2 years
  PK of IL-12-ABP as assessed by terminal half-life (t ½)
PK: CL/F of IL-12-ABP | Up to 2 years
  PK of IL-12-ABP as assessed by apparent clearance (CL/F)
PK: Vss/F of IL-12-ABP | Up to 2 years
  PK of IL-12-ABP as assessed by apparent volume of distribution at steady state (Vss/F)
Levels of ADA in serum | Up to 2 years
  Number and percentage of participants with serum levels of anti drug antibodies (ADA) after treatment
ORR by RECIST v1.1 | Up to 2 years
  Number of participants with a best overall RECIST response (BOR) of CR or PR based on RECIST v1.1
DCR by RECIST v1.1 | Up to 2 years
  Number of participants with SD, CR and PR.
DOR by RECIST v1.1 | Up to 2 years
  Time from when the criteria for RECIST v1.1 CR or PR (whichever is recorded first) was first met until the date when PD is documented
PFS by RECIST v1.1 | UP to 2 years
  Time from C1D1 to PD or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Elassal, MD, MBA, Study Director — Ankyra Therapeutics, Inc
Locations (5):
- United States (4):
  - National Cancer Institute, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Providence Cancer Institute, Portland, Oregon
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Park JC, Curti B, Butler M, Wehrenberg-Klee E, Elassal J, Tighe R, Battula S, Iodice G, Kaufman HL, Kirkwood JM. Interleukin-12 anchored drug conjugate (tolododekin alfa) in patients with advanced solid tumors: first-in-human Phase 1 trial. Nat Commun. 2025 Sep 29;16(1):8567. doi: 10.1038/s41467-025-63579-9. PMID 41022754